CLINICAL TRIAL: NCT02287298
Title: Triple Combination Therapy of Choroidal Neovascularization in Exudative Age-related Macular Degeneration - a Cost Effect and Efficient Therapeutic Treatment
Brief Title: Triple Combination Therapy of Choroidal Neovascularization in AMD, a Cost Effect and Efficient Therapeutic Treatment
Status: Completed | Type: Observational
Sponsor: The Retina Center of St. Louis County, PC (Other)
Responsible Party: Sponsor
Other Study IDs: 14-07-0540
Record Dates: First submitted 2014-09-19; First posted 2014-11-10 (Estimated); Last update posted 2016-04-06 (Estimated); Status verified 2016-04

CONDITIONS: Exudative Macular Degeneration
MeSH Terms: conditions — Wet Macular Degeneration

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 2006 TO 2010 PATIENTS: PATIENTS TREATED WITH TRIPLE COMBINATION THERAPY
  Interventions: Procedure: TRIPLE COMBINATION THERAPY
- CURRENT PATIENTS: PATIENTS TREATED WITH TRIPLE COMBINATION THERAPY AND ADDITION OF 20 MG OF ORAL ZEAXANTHIN
  Interventions: Procedure: TRIPLE COMBINATION THERAPY

INTERVENTIONS:
Procedure: TRIPLE COMBINATION THERAPY — TREATMENT WITH BEVACIZUMAB, DEXAMETHASONE AND PHOTODYNAMIC THERAPY

SUMMARY:
We propose to undertake a retrospective review of approximately 200 patients with a diagnosis of exudative macular degeneration treated with triple combination therapy (Bevacizumab, Dexamethasone and Photo-dynamic therapy) during the years of 2006 to 2010 at The Retina Center and compare those results with an additional group of approximately 200 patients also treated with triple combination therapy and 20 mg of daily oral zeaxanthin.

DETAILED DESCRIPTION:
Study parameters will include best corrected visual acuity, number of combination treatments, reduction of central foveal thickness by OCT measurement and development of exudative macular degeneration in the fellow eye. Follow up will include all patients with a minimum of two years. Retrospective review of patient charts in the office of The Retina Center.

ELIGIBILITY:
Inclusion Criteria:

- MUST HAVE AGE RELATED MACULAR DEGENERATION

Exclusion Criteria:

-

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: PATIENTS MUST HAVE A DIAGNOSIS CODE OF AGE RELATED MACULAR DEGENERATION AND MUST BE 50 YEARS OR OLDER AND HAVE EXUDATIVE AMD IN ATLEAST ONE EYE
Sampling Method: Non-Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2014-08; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
BEST CORRECTED VISUAL ACUITY | REVIEW OF EXAMINATION SHEETS

SECONDARY OUTCOMES:
NUMBER OF COMBINATION TREATMENTS | REVIEW OF CHART
REDUCTION OF CENTRAL FOVEAL THICKNESS BY OCT MEASUREMENT | REVIEW OF CHART
DEVELOPMENT OF EXUDATIVE MACULAR DEGENERATION IN THE FELLOW EYE | REVIEW OF CHART

CONTACTS AND LOCATIONS:
Overall Officials: ROBERT J OLK, MD, Principal Investigator — THE RETINA CENTER
Locations (1):
- The Retina Center, St Louis, Missouri, United States